CLINICAL TRIAL: NCT01764776
Title: A Phase I, Open Label, Multi-center, Single Dose Study to Evaluate the Pharmacokinetics of LDE225 in Healthy Subjects With Normal Hepatic Function and Subjects With Impaired Hepatic Function.
Brief Title: Effect of Hepatic Impairment on LDE225..
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDE225A2113
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2017-06

CONDITIONS: Normal Hepatic Function; Impaired Hepatic Function
Keywords: LDE225; Pharmacokinetics; PK; Postmenopausal women; normal hepatic function; mild hepatic impairment; moderate hepatic impairment; severe hepatic impairment
MeSH Terms: interventions — sonidegib

ARMS (1):
- LDE225 (Experimental): LDE225
  Interventions: Drug: LDE225

INTERVENTIONS:
Drug: LDE225 — LDE225

SUMMARY:
This study is to evaluate the pharmacokinetics and safety of 800 mg of LDE225 in subjects with impaired hepatic function and healthy subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria (all groups):

* Male and sterile or postmenopausal female age ≥18 to ≤70 years old.
* Normal Vital signs

Inclusion (group mild, moderate and severe hepatic impairment):

-Subjects with confirmed cirrhosis

Exclusion (all groups):

* Woman of childbearing potential and pregnant or lactating females or male not using condom
* Risk factors for torsades de pointes
* Clinically significant cardio-vascular disease
* severe or uncontrolled medical conditions
* Smokers consuming greater than 10 cigarettes or equivalent nicotine containing products per day.
* Use of investigational drugs (i.e. participation in any clinical investigation)

Exclusion for moderate, mild and severe groups:

* Symptoms or history of encephalopathy
* Clinical evidence of severe ascites

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
LDE225A pharmacokinetic parameter Tmax | 8 weeks
  Evaluate the pharmacokinetics of a single dose of LDE225 in subjects with impaired hepatic function as compared to healthy subjects for an 8 weeks follow up period
LDE225A pharmacokinetic parameter Cmax | 8 weeks
  Evaluate the pharmacokinetics of a single dose of LDE225 in subjects with impaired hepatic function as compared to healthy subjects for an 8 weeks follow up period
LDE225A pharmacokinetic parameter AUClast | 8 weeks
  Evaluate the pharmacokinetics of a single dose of LDE225 in subjects with impaired hepatic function as compared to healthy subjects for an 8 weeks follow up period
LDE225A pharmacokinetic parameter AUCinf | 8 weeks
  Evaluate the pharmacokinetics of a single dose of LDE225 in subjects with impaired hepatic function as compared to healthy subjects for an 8 weeks follow up period
LDE225A pharmacokinetic parameter T1/2 | 8 weeks
  Evaluate the pharmacokinetics of a single dose of LDE225 in subjects with impaired hepatic function as compared to healthy subjects for an 8 weeks follow up period

SECONDARY OUTCOMES:
Occurrence of abnormal safety laboratory parameters | 8 weeks
  Laboratory assessments
Plasma protein binding of LDE225 | 1 day
  Plasma protein binding of LDE225
Occurrence of changes in ECGs | 8 weeks
  ECGs
Occurrence of adverse event | 8 weeks
  follow up on any adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- University of Miami Div. of Clinical Pharmacology, Miami, Florida, United States
- Novartis Investigative Site, Brussels, Belgium
- Novartis Investigative Site, Sofia, Bulgaria
- Novartis Investigative Site, Berlin, Germany
- Novartis Investigative Site, Tel Aviv, Israel

REFERENCES:
- See also: Results for CLDE225A2113 from Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=14506